CLINICAL TRIAL: NCT01422863
Title: Effects of Weight Loss Through Diet and Exercise on Sleep Apnea Severity and Cardiovascular Risk in Older Adults
Brief Title: Lifestyle Interventions for Seniors With Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIZA
Record Dates: First submitted 2011-08-23; First posted 2011-08-24 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: weight loss; exercise; diet; sleep apnea; aging
MeSH Terms: conditions — Sleep Apnea, Obstructive; Weight Loss; Motor Activity; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle Intervention (Experimental)
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Participants undergo 3 months of monitored exercise, consisting of aerobic and resistance training (3 days per week for 1 hour). Participants will also meet with a registered dietician, who will prescribe an American Heart Association low fat diet. The goal is to achieve a 1-2 lb weight loss per week.

SUMMARY:
The overall goal of this study is to determine the efficacy of a lifestyle intervention, consisting of a weight loss diet and exercise on sleep apnea in older adults. The investigators will conduct a 3-month intervention in men and women who are sedentary with suspected sleep apnea. The investigators hypothesize that the intervention will lead to marked improvements in sleep apnea severity and cardiovascular risk markers.

DETAILED DESCRIPTION:
Frailty, a condition characterized by a decrease in physiological reserve and increased risk for adverse health-related outcomes, is an increased risk of aging, especially in the presence of co-morbid conditions. Sleep apnea is also highly prevalent with increasing age. Both conditions share common pathologies, suggesting that sleep apnea may increase the risk of developing or exacerbate the consequences of frailty. Lifestyle interventions as strategies for treating sleep apnea and associated co-morbidities, thereby highlighting a feasible approach by which to reduce the incidence or progression of frailty. The specific aims of this study are to: 1) determine the effectiveness of a lifestyle intervention (LI), consisting of a weight loss diet and supervised exercise, on reducing sleep apnea in older adults, and 2) determine whether this intervention is effective at improving parameters that are common to both sleep apnea and frailty, such as poor physical functional capacity and body composition, impaired or abnormal cardiometabolic function and increased levels of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* aged 60-75
* BMI between 30-42
* Apnea-Hypopnea Index above 10 events per hour (verified at baseline testing)

Exclusion Criteria:

* currently following a weight loss diet
* history of substance abuse
* participating in moderate to vigorous activity most days of the week
* history of cardiovascular disease
* currently being treated for sleep apnea
* current cigarette smoking

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Polysomnography | Baseline and 3 months
  Overnight Polysomnography will be used to measure Apnea-hypopnea index (AHI)- The number of arousals occurring over the course of the night

SECONDARY OUTCOMES:
Vascular Reactivity | Baseline and 3 months
  The Endo-PAT2000 measures endothelium-mediated changes in vascular tone using biosensors that are attached to the fingertips
maximal oxygen uptake | Baseline and 3 months
  Testing is done on a treadmill. Participants will be asked to exercise to volitional fatigue
Body composition assessment | Baseline and 3 months
  Participants will undergo Dual Energy X-ray Absorptiometry to evaluate total and regional body composition.
Muscle Strength | Baseline and 3 months
  Strength testing of the thigh will be done using an isokinetic dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Devon A Dobrosielski, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States